CLINICAL TRIAL: NCT02098044
Title: An Investigation of the Prevalence of Knee Osteoarthritis and Pain in Retired Professional Male Footballers in the United Kingdom
Brief Title: Knee Osteoarthritis Risk in Retired Professional Footballers
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Nottingham (Other)
Collaborators: Arthritis Research UK (Other); Federation Internationale de Football Association (Other); SPIRE Hospitals (Unknown); Football Association (UK) (Unknown); Professional Football Association (UK) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 13130
Record Dates: First submitted 2014-03-14; First posted 2014-03-27 (Estimated); Last update posted 2018-05-24 (Actual); Status verified 2018-05

CONDITIONS: Osteoarthritis of the Knee
Keywords: knee osteoarthritis; epidemiology; risk factors; prevalence; professional football
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Professional footballers: Retired professional footballers
- Control Population: members of the general public recruited from the east midlands region

SUMMARY:
The OA and Football Study is an epidemiological study designed to establish the prevalence of knee osteoarthritis in retired professional footballers. The study will also identify the key risk factors associated with knee osteoarthritis. The study is comprised of three phases: Phase I involves the dissemination of a questionnaire (demographic details, players history, injury and surgery and other known risk factors of OA), Phase II is a radiographic study that involves x-rays in a sample of footballers both with and without knee pain and Phase III is a case control study which will compared retired professional footballers with age-matched controls recruited from the general population in the East Midlands region.

DETAILED DESCRIPTION:
Number of Participants:

Phase I: 1000 Phase II: 855 Phase III: 500

Primary outcome: The questionnaire will contain player specific information and will include validated outcome measures such as the health status questionnaire as well as self-reported pain, recall of injury and surgery history. The results of the questionnaire will be exported firstly to Excel and subsequently, into MS Access as part of a managed database.

ELIGIBILITY:
Phase I

Inclusion Criteria:

• All current or retired professional male footballers (Registered with the Professional Footballer Association (age range 40 -80)

Phase II

Inclusion Criteria:

* Professional footballers both with and without a history of knee pain knee OA or knee surgical history
* No contraindications of the affected joint such as gout or rheumatoid arthritis
* Willingness to participate in a clinical assessment of the knee and provision of blood samples.

Phase III

Inclusion Criteria for controls:

* Over the age of 40 (age range 40 - 80)
* Both with and without a history of knee pain over at least the last 1 year
* No history of significant trauma, injury or surgery to the lower limb
* American College of Rheumatology (ACR) classification of OA based on physical examination and clinical presentation: Pain in the knee and three of the following; over the age of 50, less than 30 minutes of morning stiffness, crepitus on active motion, bony tenderness, bony enlargement and no palpable warmth of synovium.

Phase I

Exclusion Criteria:

* Not a registered professional footballer (current or past)
* Inaccurate information (discrepancy with questionnaire information compared to other football records. This will be verified by the co-investigator, Dr Fernandes and Mr Sanjay Parekh)
* Incomplete questionnaire or duplicate questionnaire.

Phase II

Exclusion Criteria:

* Not a registered professional footballer
* No written informed consent to participate

Phase III

Exclusion Criteria:

* Aged 39 and under
* Comorbidities such as rheumatoid arthritis, gout, osteoporosis
* History of injury, trauma or surgery to the lower limb.

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Retired footballers will be recruited from a database of retired professional footballers. (cases)
  The members of the general public will be recruited from the general population in the East Midlands region. (controls)
Sampling Method: Probability Sample
Enrollment: 1300 (Actual)
Dates: Start 2014-11; Primary Completion 2016-01 (Actual); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Self Reported Knee Pain | up to 12 months
  Questionnaire data with regards to acute knee pain, type of pain, duration of pain and knee injury and knee surgery history.

SECONDARY OUTCOMES:
Radiographic Knee OA changes | up to 12 months
  Bilateral x rays using standardised rigs for 2 views. Postero-anterior view (30 degrees flexion, weight bearing) and skyline views.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Doherty, MD, Principal Investigator — University of Nottingham
Locations (1):
- Academic Rheumatology, Nottingham, Nottinghamshire, United Kingdom

REFERENCES:
- [Background] Drawer S, Fuller CW. Evaluating the level of injury in English professional football using a risk based assessment process. Br J Sports Med. 2002 Dec;36(6):446-51. doi: 10.1136/bjsm.36.6.446. PMID 12453840
- [Background] Zhang W, McWilliams DF, Ingham SL, Doherty SA, Muthuri S, Muir KR, Doherty M. Nottingham knee osteoarthritis risk prediction models. Ann Rheum Dis. 2011 Sep;70(9):1599-604. doi: 10.1136/ard.2011.149807. Epub 2011 May 25. PMID 21613308
- [Derived] Fernandes GS, Parekh SM, Moses J, Fuller CW, Scammell B, Batt ME, Zhang W, Doherty M. Depressive symptoms and the general health of retired professional footballers compared with the general population in the UK: a case-control study. BMJ Open. 2019 Sep 8;9(9):e030056. doi: 10.1136/bmjopen-2019-030056. PMID 31501119